CLINICAL TRIAL: NCT03691727
Title: A Phase 1/2a Exploratory Clinical Trial: Induced Suppression of Platelets Activity in Aneurysmal SAH Management (iSPASM)
Brief Title: Induced Suppression of Platelets Activity in Aneurysmal SAH Management (iSPASM)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David Hasan (Other)
Responsible Party: Sponsor-Investigator, David Hasan, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201805823
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Results first posted 2021-10-04 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2020-08

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Tirofiban; Neurologic Examination; Surveys and Questionnaires; Vital Signs

STUDY DESIGN:
Intervention Model Description: All subjects will be randomized 2:1, Aggrastat vs. placebo.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- tirofiban hydrochloride (AGGRASTAT®) (Experimental): tirofiban hydrochloride (AGGRASTAT®) administered continuously over the course of 7 days.
  MRI Neurological Exam Vital Signs Questionnaires
  Interventions: Drug: tirofiban hydrochloride (AGGRASTAT®); Diagnostic Test: MRI; Diagnostic Test: Neurological Exam; Behavioral: Questionnaires; Diagnostic Test: Vital Signs
- Standard of Care Control Arm (Active Comparator): Standard of Care Treatment MRI Neurological Exam Vital Signs Questionnaires
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Neurological Exam; Behavioral: Questionnaires; Diagnostic Test: Vital Signs; Other: Standard of Care Treatment

INTERVENTIONS:
Drug: tirofiban hydrochloride (AGGRASTAT®) — Participants will have intravenous Aggrastat administered continuously over the course of 7 days in the setting of subarachnoid hemorrhage at least 12 hours post clinically indicated Endovascular Coil Embolization procedure.
  Arms: tirofiban hydrochloride (AGGRASTAT®)
Diagnostic Test: MRI — Participants will undergo 2 MRIs administered within 24 hours post Coil Embolization procedure and prior to discharge to monitor for ischemic changes.
Diagnostic Test: Neurological Exam — Neurological exams will be done at screening, randomization, days 2-7, discharge, 6 week, 6 month, and one year follow up visits.
Behavioral: Questionnaires — Quality of Life in Brain Injury - Overall Scale (QOLIBRI-OS) and the Lawton Instrumental Activities of Daily Living (IADL) will be administered at 6 month and 1 year follow up visits.
Diagnostic Test: Vital Signs — Vital signs which include temperature, respiration rate, blood pressure and O2 stats will be done at screening, randomization, days 2-7, discharge, 6 week, 6 month, and one year follow up visits.
Other: Standard of Care Treatment — Participants will receive standard of care treatment and will not receive study drug.
  Arms: Standard of Care Control Arm

SUMMARY:
This is a phase 1/2a, randomized, double blind, single-center study comparing standard care alone to standard care with Aggrastat in patients diagnosed with aneurysmal subarachnoid hemorrhage.

DETAILED DESCRIPTION:
This is a phase 1/2a, randomized, double blind, single-center study comparing standard care alone to standard care with Aggrastat in patients diagnosed with aneurysmal subarachnoid hemorrhage. The investigational plan is to explore the safety profile of Aggrastat administered continuously over 7 days, beginning at least 12 hours after a clinically indicated Endovascular Coil Embolization procedure.

As a part of the study, qualifying subjects will undergo two MRI scans, one at baseline and again prior to discharge. A neurological exam and vital signs will be administered at baseline, daily during drug administration, and at follow-up visits. Additional assessments include administration of the following questionnaires: mRS score, IADL, and QOLIBRI-OS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 85 years
* Hunt and Hess scale ≤ 4 at time of admission or following EVD placement.
* CT showing modified Fisher grade 1-4 aSAH on admission.
* The Modified Fisher CT rating scale: Grade 1 (minimal or diffuse thing SAH without IVH); Grade 2 (minimal or thin SAH with IVH), Grade 3 (thick cisternal clot without IVH), Grade 4 (thick cisternal clot with IVH)
* Placement of EVD on admission.
* Diagnosis of aSAH occurred < 24 hours prior to presentation at the treating facility.
* Initiation of aneurysm securement procedure occurred ≤ 24 hours from admission to the treating facility.
* All aneurysm(s) suspected to be responsible for the hemorrhage or potentially responsible for the hemorrhage must be secured in the following manner prior to enrollment: Endovascular Coil Embolization with a post-embolization Raymond-Roy Score of 1 (Complete) or 2 (Residual Neck)
* Ability to screen the patient and obtain head CT, CT perfusion, and CCTA on admission, a head CT following EVD placement, during EVD weaning period and following VP shunt placement.
* No evidence of a significant new focal neurological deficit after the angiogram, including monoparesis / monoplegia, hemiparesis / hemiplegia, or receptive, expressive, or global aphasia. Minor cranial nerve defect without any other new findings is permissible. The treating physician should use their best clinical judgement as to whether a significant neurological decline has occurred due to the procedure.
* Patient or their Legally Authorized Representative (LAR) has provided written informed consent.

Exclusion Criteria:

* Angio-negative SAH, defined as a subarachnoid hemorrhage with an angiogram that does not show a related intracranial hemorrhage.
* A likely hemorrhage event preceding the ictus due to the increased risk of early vasospasm. Prior sentinel headache with negative CT or prior sentinel headache where the patient did not seek medical attention does not exclude the patient.
* Surgical clipping of the ruptured aneurysm or any non-ruptured aneurysm on the same admission prior to enrollment.
* SAH not caused by aneurysm rupture or aneurysm is identified to be traumatic, mycotic, blister or fusiform type by catheter angiography.
* Any intracranial stent placement or non-coil intra-aneurysmal device (i.e., stent- assisted coiling with Neuroform, Enterprise, LVIS, LVIS Jr, Barrel Stent, Pulse Rider, LUNA, Medina or a similar device) where the stent device is implanted to treat the ruptured aneurysm.
* A medical diagnosis that requires continuous use of clopidogrel, ticagrelor, or tirofiban during study drug infusion.
* Antiplatelet therapy using clopidogrel, ticagrelor or tirofiban during the endovascular procedure that continues > 24 post embolization.
* Multiple aneurysms that may have been untreated and a potential etiology for rupture.
* Femoral arteriotomy stick above the inferior epigastric artery OR angiographic, CT, or clinical evidence of an arteriotomy related retroperitoneal hematoma or large flank hematoma. A stable groin hematoma is not an exclusion.
* Thrombocytopenia (platelet count less than 100,000 - assuming clumping has been ruled out as a cause), confirmed active disseminated intravascular coagulation (DIC) at the time of enrollment OR a documented history of coagulopathy or bleeding diathesis.
* New parenchymal hemorrhage or new infarction larger the 15cc in volume (clinically significant), or worsening midline shift as seen on the post-coiling, pre-enrollment head CT when compared to baseline admission head CT. New hyperdensity on CT scan related to contrast staining is not an exclusion.
* Patient developed SAH-induced cardiac stunning prior to enrollment, with an ejection fraction < 40%.
* Thrombolytic therapy within 24 hours prior to enrollment (rtPA, urokinase, etc.)
* Concurrent significant intracranial pathology identified prior to enrollment, including but not limited to, Moyamoya disease, high suspicion or documented CNS vasculitis, severe fibromuscular dysplasia, arteriovenous malformation, arteriovenous fistula, significant cervical or intracranial atherosclerotic stenotic disease ≥ 70%, or malignant brain tumor.
* Known seizure or epilepsy disorder (diagnosed prior to this aSAH diagnosis) where anti-epileptic medication was previously taken by the patient or have been recommended to be taken by the patient. Childhood seizures that have resolved and no longer require treatment are not part of this exclusion criteria.
* Serious co-morbidities that could confound study results including but not limited to: Multiple Sclerosis, dementia, severe major depression, cancer likely to cause death in 2 years, multi-system organ failure, or any other conditions that could cause any degree of cognitive impairment.
* Immunosuppression therapy including chronic corticosteroid usage.
* Remote history of previous ruptured cerebral aneurysm.
* History of gastrointestinal hemorrhage or major systemic hemorrhage within 30 days, hemoglobin less than 8 g/dL, INR ≥ 1.5, severe liver impairment defined as AST, ALT, AP, GGT > 2 x normal.
* Creatinine clearance < 30 mL/min.
* Major surgery within 30 days with contraindication to antiplatelet therapy.
* Currently pregnant.
* Contraindication for MRI
* Contraindication to antiplatelet tirofiban:

  1. active internal bleeding or a history of bleeding diathesis within the previous 30 days
  2. A history of thrombocytopenia following prior exposure to AGGRASTAT
  3. history, symptoms, or findings suggestive of aortic dissection
  4. acute pericarditis
* Actual Body Weight > 150 kg (due to the lack of safety data)
* 2 or more passes for the ventricular catheter at time of placement.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zanaty M, Allan L, Samaniego EA, Piscopo A, Ryan E, Torner JC, Hasan D. Phase 1/2a Trial of ISPASM. Stroke. 2021 Dec;52(12):3750-3758. doi: 10.1161/STROKEAHA.121.034578. Epub 2021 Sep 2. PMID 34470496

RESULTS

PARTICIPANT FLOW:
Groups:
- Tirofiban Hydrochloride (AGGRASTAT®): tirofiban hydrochloride (AGGRASTAT®) administered continuously over the course of 7 days.
  MRI Neurological Exam Vital Signs Questionnaires
  tirofiban hydrochloride (AGGRASTAT®): Participants will have intravenous Aggrastat administered continuously over the course of 7 days in the setting of subarachnoid hemorrhage at least 12 hours post clinically indicated Endovascular Coil Embolization procedure.
  MRI: Participants will undergo 2 MRIs administered within 24 hours post Coil Embolization procedure and prior to discharge to monitor for ischemic changes.
  Neurological Exam: Neurological exams will be done at screening, randomization, days 2-7, discharge, 6 week, 6 month, and one year follow up visits.
  Questionnaires: Quality of Life in Brain Injury - Overall Scale (QOLIBRI-OS) and the Lawton Instrumental Activities of Daily Living (IADL) will be administered at 6 month and 1 year follow up visits.
  Vital Signs: Vital signs which include temperature, respiration rate, blood pressure and O2 stats will be done at screening, randomization, days 2-7, discharge, 6 week, 6 month, and one year follow up visits.
Period: Overall Study
Arm/Group | Tirofiban Hydrochloride (AGGRASTAT®) | Standard of Care Control Arm
Started | 18 | 12
Completed | 16 | 11
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tirofiban Hydrochloride (AGGRASTAT®) | Standard of Care Control Arm | Total
Number analyzed (Participants) | 18 | 12 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 25
  >=65 years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 6 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 13 | 9 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Intracranial Hemorrhage (Symptomatic and Asymptomatic)
Description: The hypothesis is that the prevalence of intracranial hemorrhage (symptomatic and asymptomatic) secondary to ventriculostomy/VPS placement during the course of Aggrastat use is within 10% difference when compared to control using Day 1 and Day 7 non-contrast head CT to determine.
Time Frame: Day 1 to Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Tirofiban Hydrochloride (AGGRASTAT®) | Standard of Care Control Arm
Number analyzed (Participants) | 18 | 12
Participants | 2 | 1

2. Primary Outcome: Number of Participants With Delayed Cerebral Ischemia /Clinical Vasospasm
Description: The measurement of then incidence of delayed cerebral ischemia /clinical vasospasm in Tirofiban/Aggrastat group vs. placebo
Time Frame: Day 1 to Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Tirofiban Hydrochloride (AGGRASTAT®) | Standard of Care Control Arm
Number analyzed (Participants) | 18 | 12
Participants | 1 | 4

ADVERSE EVENTS:
Time Frame: Enrollment to 1 year follow up appointment (+/- 1 month from enrollment)
Description: All adverse events were collected for 11 days after initial dose. From Day 11 until 6 weeks serious adverse events and adverse events of special interest were monitored. From 6 weeks until 1 year follow up appointment only serious adverse events were monitored.
Arm/Group | Tirofiban Hydrochloride (AGGRASTAT®) | Standard of Care Control Arm
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/12
Serious Adverse Events (participants affected / at risk) | 18/18 | 12/12
Other Adverse Events (participants affected / at risk) | 18/18 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tirofiban Hydrochloride (AGGRASTAT®) (N=18) | Standard of Care Control Arm (N=12)
Acute Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cerebral Edema (Nervous system disorders) | 1 | 0
Clinical Vasospasm (Nervous system disorders) | 1 | 4
Deep Vein Thrombosis (DVT) (Vascular disorders) | 1 | 2
External Ventricular Drain (EVD) Malfunction (Product Issues) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Ventriculitis (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Enterocolitis Infectious (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 2 | 0
Frontal Lobe Ischemia (Nervous system disorders) | 0 | 1
Hypotension (Cardiac disorders) | 4 | 0
Ileus (Nervous system disorders) | 0 | 1
Intracranial Hypertension (Nervous system disorders) | 0 | 1
Intracranial Hypertension with Cerebral Edema (Nervous system disorders) | 1 | 0
Neurogenic Pulmonary Edema (Nervous system disorders) | 1 | 0
Parietal Punctate Infarcts (Nervous system disorders) | 1 | 0
Radiographic Vasospasm (Nervous system disorders) | 2 | 0
Subdural Hematoma (Nervous system disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Vasogenic Edema (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tirofiban Hydrochloride (AGGRASTAT®) (N=18) | Standard of Care Control Arm (N=12)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1
External Ventricular Drain Malfunction (Product Issues) | 1 | 0
Fever (Infections and infestations) | 13 | 9
Headache (Nervous system disorders) | 4 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Acute Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Agitation (Psychiatric disorders) | 4 | 0
Altered Mental Status (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Urinary Tract Infection (UTI) (Immune system disorders) | 2 | 0
Back Pain (General disorders) | 0 | 2
Bigeminy (Cardiac disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 3
Polyuria (Renal and urinary disorders) | 9 | 6
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1
Delirium (Psychiatric disorders) | 4 | 4
Diarrhea (Metabolism and nutrition disorders) | 3 | 5
Dysphagia (Gastrointestinal disorders) | 3 | 0
Cerebral Salt Wasting Phenomenon (Nervous system disorders) | 4 | 1
Dysphasia (General disorders) | 0 | 1
Electrocardiogram (EKG) Changes (Cardiac disorders) | 2 | 0
Ear Pain (General disorders) | 1 | 0
Flank Pain (General disorders) | 1 | 0
Groin Yeast Infection (Infections and infestations) | 1 | 0
High Glucose Level (Endocrine disorders) | 1 | 0
High Platelet Count (Blood and lymphatic system disorders) | 8 | 3
High White Blood Cell (WBC) Count (Blood and lymphatic system disorders) | 11 | 6
Hip Pain (General disorders) | 2 | 0
Hypertension (Cardiac disorders) | 2 | 0
Hypervolemia (Blood and lymphatic system disorders) | 0 | 1
Intravenous Line (IV) Infiltration (Surgical and medical procedures) | 0 | 1
Incontinence (Gastrointestinal disorders) | 1 | 0
Leg Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Low Creatinine Level (Renal and urinary disorders) | 7 | 6
Low Hematocrit (Blood and lymphatic system disorders) | 10 | 8
Low Hemoglobin (Blood and lymphatic system disorders) | 12 | 8
Low Potassium (Renal and urinary disorders) | 12 | 11
Low Sodium (Renal and urinary disorders) | 12 | 5
Nausea (Gastrointestinal disorders) | 3 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pericatheter Right Frontal Hypodensity (Nervous system disorders) | 1 | 0
Periorbital Pain (Eye disorders) | 1 | 0
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Somnolence (Nervous system disorders) | 3 | 0
Tachycardia (Cardiac disorders) | 5 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Urinary Retention (Renal and urinary disorders) | 6 | 0
Vaginal Yeast Infection (Infections and infestations) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT03691727/Prot_SAP_000.pdf